CLINICAL TRIAL: NCT00842751
Title: Pharmacokinetics of a Novel Oral Testosterone Undecanoate Formulation With Concomitant Inhibition of 5alpha-Reductase by Finasteride
Brief Title: Oral T7 Oral Testosterone in Man
Acronym: Oral T7
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Amory, Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 35724-W; 1K23HD045386 (NIH); 5U54HD042454 (NIH)
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Males; Male Contraceptive
Keywords: 5α-reductase; androgen; dihydrotestosterone (DHT); drug delivery; oestradiol
MeSH Terms: interventions — Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Testosterone Undecanoate + placebo finasteride (Placebo Comparator): Acyline 300mcg/kg subcutaneous on days 1, 15 and 29 + Testosterone Undecanoate (TU)200mg twice daily, orally for 7 days + placebo finasteride twice daily, orally for 7 days during one of the three intervention periods (First Intervention, Second Intervention or Third Intervention)
  Interventions: Drug: First Intervention (7 days); Other: First Washout (7 days)
- Testosterone Undecanoate + Finasteride 0.5mg (Experimental): Acyline 300mcg/kg subcutaneous on days 1, 15 & 29 + testosterone undecanoate 200mg, twice daily orally for 7 days + finasteride 0.5mg twice daily, orally for 7 days during one of the three intervention periods (First Intervention, Second Intervention or Third Intervention)
  Interventions: Drug: Second Intervention (7 days); Other: Second wash-out period
- Testosterone Undecanoate + Finasteride 1mg (Experimental): Acyline 300mcg/kg subcutaneous on days 1, 15 & 29 + testosterone undecanoate 200mg, twice daily orally for 7 days + finasteride 1mg twice daily, orally for 7 days during one of the three intervention periods ((First Intervention, Second Intervention or Third Intervention)
  Interventions: Drug: Third Intervention (7 days)

INTERVENTIONS:
Drug: First Intervention (7 days) — Acyline 300mcg/kg subcutaneous (days 1, 15 & 29) + testosterone undecanoate 200 mg, twice daily orally + finasteride placebo
  Other Names: propecia
  Arms: Testosterone Undecanoate + placebo finasteride
Other: First Washout (7 days) — Washout of 7 days between each of the 3 treatment arms
  Other Names: no active drugs
  Arms: Testosterone Undecanoate + placebo finasteride
Drug: Second Intervention (7 days) — Acyline 300mcg/kg subcutaneous + testosterone undecanoate 200 mg, twice daily orally + finasteride 0.5mg twice daily, orally
  Other Names: propecia
  Arms: Testosterone Undecanoate + Finasteride 0.5mg
Drug: Third Intervention (7 days) — Acyline 300mcg/kg subcutaneous + testosterone undecanoate 200 mg, twice daily orally + finasteride 1mg twice daily, orally
  Other Names: propecia
  Arms: Testosterone Undecanoate + Finasteride 1mg
Other: Second wash-out period — Washout of 7 days between each of the 3 treatment arms
  Other Names: no active drug
  Arms: Testosterone Undecanoate + Finasteride 0.5mg

SUMMARY:
The purpose of this study is to test how the body absorbs and processes new forms of oral testosterone. Information gained during the study may help develop better forms of testosterone therapy in the future.

DETAILED DESCRIPTION:
We will be using three drugs: The first, acyline, temporarily turns off the body's production of testosterone for about two weeks. Subjects will receive acyline as shots three times over a six-week drug administration period. During the time when the body's production of testosterone is turned off, we will give testosterone either by itself or with a medication called finasteride by mouth twice daily for one week to see how much is absorbed and present in the bloodstream after administration. Subjects will go through three one-week study drug exposure periods. During two of the three one-week study drug administration periods subjects will also take a second medication, finasteride, by mouth twice daily. On the last day of each one-week drug administration period, subjects will be admitted to the University of Washington General Clinical Research Center overnight for monitoring of your blood testosterone levels. There will be 3 overnight visits for this study. This study will allow us to determine the absorption of testosterone taken by mouth, and the relative impact of two different doses of oral finasteride on testosterone absorption.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 50 years of age
* In good health based on normal screening evaluation (consisting of a medical history, physical exam normal serum chemistry, hematology, and baseline hormone levels.
* Must agree to not participate in another research drug study
* Must agree to not donate blood
* Must be willing to comply with the study protocol and procedures

Exclusion Criteria:

* Men in poor general health, with abnormal blood results (clinical laboratory tests or hormone values)
* A known history of alcohol or drug abuse
* Participation in a long-term male contraceptive study within the past month
* History of bleeding disorders or current use of anti-coagulants
* History of sleep apnea
* History of major psychiatric disorder
* Body mass index > 37
* Infertility
* Hematocrit > 55 or < 30
* PSA >4

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Amory, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Katznelson L, Finkelstein JS, Schoenfeld DA, Rosenthal DI, Anderson EJ, Klibanski A. Increase in bone density and lean body mass during testosterone administration in men with acquired hypogonadism. J Clin Endocrinol Metab. 1996 Dec;81(12):4358-65. doi: 10.1210/jcem.81.12.8954042.
- [Background] Behre HM, Kliesch S, Leifke E, Link TM, Nieschlag E. Long-term effect of testosterone therapy on bone mineral density in hypogonadal men. J Clin Endocrinol Metab. 1997 Aug;82(8):2386-90. doi: 10.1210/jcem.82.8.4163. PMID 9253305
- [Background] Bhasin S, Bremner WJ. Clinical review 85: Emerging issues in androgen replacement therapy. J Clin Endocrinol Metab. 1997 Jan;82(1):3-8. doi: 10.1210/jcem.82.1.3640. No abstract available. PMID 8989221
- [Background] Wang C, Alexander G, Berman N, Salehian B, Davidson T, McDonald V, Steiner B, Hull L, Callegari C, Swerdloff RS. Testosterone replacement therapy improves mood in hypogonadal men--a clinical research center study. J Clin Endocrinol Metab. 1996 Oct;81(10):3578-83. doi: 10.1210/jcem.81.10.8855804.
- [Background] Snyder PJ, Peachey H, Berlin JA, Hannoush P, Haddad G, Dlewati A, Santanna J, Loh L, Lenrow DA, Holmes JH, Kapoor SC, Atkinson LE, Strom BL. Effects of testosterone replacement in hypogonadal men. J Clin Endocrinol Metab. 2000 Aug;85(8):2670-7. doi: 10.1210/jcem.85.8.6731. PMID 10946864
- [Background] Kelch RP, Jenner MR, Weinstein R, Kaplan SL, Grumbach MM. Estradiol and testosterone secretion by human, simian, and canine testes, in males with hypogonadism and in male pseudohermaphrodites with the feminizing testes syndrome. J Clin Invest. 1972 Apr;51(4):824-30. doi: 10.1172/JCI106877. PMID 4259253
- [Background] Weinstein RL, Kelch RP, Jenner MR, Kaplan SL, Grumbach MM. Secretion of unconjugated androgens and estrogens by the normal and abnormal human testis before and after human chorionic gonadotropin. J Clin Invest. 1974 Jan;53(1):1-6. doi: 10.1172/JCI107526. PMID 4271572
- [Background] Bagatell CJ, Bremner WJ. Androgens in men--uses and abuses. N Engl J Med. 1996 Mar 14;334(11):707-14. doi: 10.1056/NEJM199603143341107. No abstract available. PMID 8594431
- [Background] Fossa SD, Opjordsmoen S, Haug E. Androgen replacement and quality of life in patients treated for bilateral testicular cancer. Eur J Cancer. 1999 Aug;35(8):1220-5. doi: 10.1016/s0959-8049(99)00123-9. PMID 10615233
- [Background] Amory JK, Matsumoto AM. The therapeutic potential of testosterone patches. Expert Opin Investig Drugs. 1998 Dec;7(12):1977-85. doi: 10.1517/13543784.7.12.1977. PMID 15991940
- [Background] Swerdloff RS, Wang C, Cunningham G, Dobs A, Iranmanesh A, Matsumoto AM, Snyder PJ, Weber T, Longstreth J, Berman N. Long-term pharmacokinetics of transdermal testosterone gel in hypogonadal men. J Clin Endocrinol Metab. 2000 Dec;85(12):4500-10. doi: 10.1210/jcem.85.12.7045. PMID 11134099
- [Background] Nieschlag E, Mauss J, Coert A, Kicovic P. Plasma androgen levels in men after oral administration of testosterone or testosterone undecanoate. Acta Endocrinol (Copenh). 1975 Jun;79(2):366-74. doi: 10.1530/acta.0.0790366. PMID 1173495
- [Background] Johnsen SG, Bennett EP, Jensen VG. Therapeutic effectiveness of oral testosterone. Lancet. 1974 Dec 21;2(7895):1473-5. doi: 10.1016/s0140-6736(74)90216-5. No abstract available. PMID 4140393
- [Background] Daggett PR, Wheeler MJ, Nabarro JD. Oral testosterone, a reappraisal. Horm Res. 1978;9(3):121-9. doi: 10.1159/000178904. PMID 640576
- [Background] Amory JK, Bremner WJ. Oral testosterone in oil plus dutasteride in men: a pharmacokinetic study. J Clin Endocrinol Metab. 2005 May;90(5):2610-7. doi: 10.1210/jc.2004-1221. Epub 2005 Feb 15. PMID 15713724
- [Background] Amory JK, Page ST, Bremner WJ. Oral testosterone in oil: pharmacokinetic effects of 5alpha reduction by finasteride or dutasteride and food intake in men. J Androl. 2006 Jan-Feb;27(1):72-8. doi: 10.2164/jandrol.05058. PMID 16400081
- [Background] Amory JK, Watts NB, Easley KA, Sutton PR, Anawalt BD, Matsumoto AM, Bremner WJ, Tenover JL. Exogenous testosterone or testosterone with finasteride increases bone mineral density in older men with low serum testosterone. J Clin Endocrinol Metab. 2004 Feb;89(2):503-10. doi: 10.1210/jc.2003-031110. PMID 14764753
- [Background] Herbst KL, Coviello AD, Page S, Amory JK, Anawalt BD, Bremner WJ. A single dose of the potent gonadotropin-releasing hormone antagonist acyline suppresses gonadotropins and testosterone for 2 weeks in healthy young men. J Clin Endocrinol Metab. 2004 Dec;89(12):5959-65. doi: 10.1210/jc.2003-032123. PMID 15579744
- [Background] Amory JK, Wang C, Swerdloff RS, Anawalt BD, Matsumoto AM, Bremner WJ, Walker SE, Haberer LJ, Clark RV. The effect of 5alpha-reductase inhibition with dutasteride and finasteride on semen parameters and serum hormones in healthy men. J Clin Endocrinol Metab. 2007 May;92(5):1659-65. doi: 10.1210/jc.2006-2203. Epub 2007 Feb 13. PMID 17299062
- [Result] Roth MY, Dudley RE, Hull L, Leung A, Christenson P, Wang C, Swerdloff R, Amory JK. Steady-state pharmacokinetics of oral testosterone undecanoate with concomitant inhibition of 5alpha-reductase by finasteride. Int J Androl. 2011 Dec;34(6 Pt 1):541-7. doi: 10.1111/j.1365-2605.2010.01120.x. Epub 2010 Oct 24. PMID 20969601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men age 18-52 in good health were recruited through local newspapers and college campus flyers.
Pre-assignment Details: 12 subjects were screened; 11 enrolled (1 did not meet inclusion criteria-abnormal liver function test at baseline and excessive alcohol use). Each subject was administered each of the three treatments over a 6-week period with 1 week of no treatment (wash-out) between each of the treatment period.
Groups:
- Acyline + Testosterone Undecanoate + Placebo Finasteride: Acyline 300 mcg/kg +Testosterone Undecanoate 200 mg, BID orally + placebo finasteride
Period: Overall Study
Arm/Group | Acyline + Testosterone Undecanoate + Placebo Finasteride
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Each subject was administered each of the three treatments over a 6-week period with 1 week of no treatment (wash-out) between each of the treatment period.
Arm/Group | All Study Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Weight [Mean (Standard Deviation); unit: kg] | 80 (13)
Height [Mean (Standard Deviation); unit: cm] | 181 (7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 24 (3)
Serum testosterone concentration [Mean (Standard Deviation); unit: ng/dL] | 405 (14)
Serum dihydrotestosterone concentration [Mean (Standard Deviation); unit: ng/dL] | 32 (12)
Serum oestradiol concentration [Median (Standard Deviation); unit: pg/mL] | 15 (5)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Testosterone Concentration
Description: Area under the curve of serum testosterone Pharmacokinetic measures time-weighted mean concentration calculated as area under the concentration curve (AUC) divided by time from initiation of dosing for the morning dose and corrected for differences in baseline hormone concentration.
Time Frame: 0,1,2,4,8,and 12-hour post dose
Population: All participant received all treatments and is, therefore, included in the analysis population for all groups.
Measure: Geometric Mean (Inter-Quartile Range); unit: ng*hr/dL
Groups:
- Acyline +Testosterone Undecanoate + Placebo: Acyline 300 mcg/kg SC +Testosterone Undecanoate 200 mg, BID orally + Placebo Finasteride
- Acyline +Testosterone Undecanoate + 0.5mg Finasteride: Acyline 300 mcg/kg SC + Testosterone Undecanoate 200 mg, BID orally + Finasteride 0.5 mg, BID orally
- Acyline +Testosterone Undecanoate + 1mg Finasteride: Acyline 300 mcg/kg SC + Testosterone Undecanoate 200 mg, BID orally + Finasteride 1 mg, BID orally
Arm/Group | Acyline +Testosterone Undecanoate + Placebo | Acyline +Testosterone Undecanoate + 0.5mg Finasteride | Acyline +Testosterone Undecanoate + 1mg Finasteride
Number analyzed (Participants) | 11 | 11 | 11
ng*hr/dL | 471 [381 to 581] | 444 [358 to 551] | 543 [439 to 671]

2. Primary Outcome: Serum Dihydrotestosterone Concentration
Description: Area under the curve of serum dihydrotestosterone
Time Frame: 0,1,2,4,8,and 12-hour post dose
Population: All participants received all treatment, and is therefore, included in the analysis population for all three treatment groups.
Measure: Geometric Mean (Inter-Quartile Range); unit: ng*hr/dL
Groups:
- Acyline +Testosterone Undecanoate + Placebo: Acyline 300 mcg/kg subcutaneous (SC) +Testosterone Undecanoate 200 mg, BID orally + Placebo finasteride
- Acyline + Testosterone Undecanoate + 0.5mg Finasteride: Acyline 300 mcg/kg SC +Testosterone Undecanoate 200 mg, BID orally + 0.5mg finasteride
- Acyline + Testosterone Undecanoate + 1mg Finasteride: Acyline 300 mcg/kg SC +Testosterone Undecanoate 200 mg, BID orally + 1mg finasteride
Arm/Group | Acyline +Testosterone Undecanoate + Placebo | Acyline + Testosterone Undecanoate + 0.5mg Finasteride | Acyline + Testosterone Undecanoate + 1mg Finasteride
Number analyzed (Participants) | 11 | 11 | 11
ng*hr/dL | 154 [125 to 190] | 118 [96 to 146] | 125 [102 to 154]

3. Primary Outcome: Serum Estradiol Concentration
Description: Area under the curve of serum estradiol
Time Frame: 0,1,2,4,8,and 12-hour post dose
Population: as for outcome 2
Measure: Geometric Mean (Inter-Quartile Range); unit: ng*hr/dL
Groups:
- Acyline +Testosterone Undecanoate + Placebo: Acyline 300 mcg/kg SC + Testosterone Undecanoate 200 mg, twice daily (BID) orally + placebo finasteride
- Acyline +Testosterone Undecanoate + 1mg Finasteride: Acyline 300 mcg/kg SC +Testosterone Undecanoate 200 mg, BID orally + 1mg finasteride
Arm/Group | Acyline +Testosterone Undecanoate + Placebo | Acyline + Testosterone Undecanoate + 0.5mg Finasteride | Acyline +Testosterone Undecanoate + 1mg Finasteride
Number analyzed (Participants) | 11 | 11 | 11
ng*hr/dL | 7.9 [6.4 to 9.7] | 6.5 [5.2 to 8.0] | 7.2 [5.8 to 8.9]

ADVERSE EVENTS:
Groups:
- First Intervention: Acyline 300mcg/kg subcutaneous on days 1, 15 & 29 + Testosterone Undecanoate 200 mg, twice daily, orally + Finasteride placebo, twice daily, orally
- Second Intervention: Acyline 300mcg/kg subcutaneous on days 1, 15 & 29 + Testosterone Undecanoate 200 mg, BID orally + Finasteride 0.5mg, twice a day, orally
- Third Intervention: Acyline 300mcg/kg subcutaneous on days 1, 15 & 29 + Testosterone Undecanoate 200 mg, twice daily orally + Finasteride 1mg, twice a day, orally
Arm/Group | First Intervention | Second Intervention | Third Intervention
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 4/11 | 2/11 | 3/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Intervention (N=11) | Second Intervention (N=11) | Third Intervention (N=11)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Testicular Pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Upset Stomach & Reflux (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes